CLINICAL TRIAL: NCT03395886
Title: Remifentanil Versus Dexmedetomidine for Post-Cardiac Surgery Patients With Noninvasive Ventilation Intolerance: A Prospective, Observational,Cohort Study
Brief Title: Remifentanil Versus Dexmedetomidine for Post-Cardiac Surgery Patients With Noninvasive Ventilation Intolerance
Acronym: REDNIVIN
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REDNIVIN
Record Dates: First submitted 2017-12-21; First posted 2018-01-10 (Actual); Results first posted 2019-11-29 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-08

CONDITIONS: Cardiac Surgery
Keywords: noninvasive ventilation; remifentanil; dexmedetomidine; cardiac surgery
MeSH Terms: interventions — Remifentanil; Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- remifentanil group: Eligible patients will receive a continuous infusion of remifentanil starting with 0.05 μg/kg/min. The doses will be adjusted according to the sedation satisfaction (sedation target is to achieve NIV-intolerance score 1-2), and the maximum dose is 0.12 μg/kg/min.
  Interventions: Drug: Remifentanil
- dexmedetomidine group: Eligible patients will receive a continuous infusion of dexmiditomidine starting with 0.5 μg/kg/h. The doses will be adjusted according to the sedation satisfaction (sedation target is to achieve NIV-intolerance score 1-2), and the maximum dose is 1 μg/kg/h.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Remifentanil — The noninvasive ventilation intolerated patients was sedated by remifentanil.
  Groups: remifentanil group
Drug: Dexmedetomidine — The noninvasive ventilation intolerated patients was sedated by dexmeditomidine.
  Groups: dexmedetomidine group

SUMMARY:
The aim of this study is to compare the sedation effects between remifentanil and dexmedetomidine in post-cardiac surgical patients who developed noninvasive ventilation (NIV) intolerance.

DETAILED DESCRIPTION:
This study is a prospective,observational,cohort study. Data of post-cardiac surgical patients who receives noninvasive ventilation (NIV) in the investigators' cardiac surgical intensive care unit are prospectively collected into a database for further analyzation since January 2018. Tolerance of NIV is estimated by a four-point NIV intolerance score system: A score of 1 indicates a comfortable and relaxed patient tolerating NIV; a score of 2 indicates mild intolerance with some discomfort and occasional grabbing at the NIV mask; a score of 3 indicates moderate intolerance and discomfort with the NIV mask most of the time with frequent grabbing at the mask (sometimes pulling it off); and a score of 4 indicates severe NIV intolerance with agitation or/and an inability to leave the NIV mask in place. Participants who receives re-intubation will be recorded as 4 points. Application of remifentanil or dexmedetomidine will be initiated when a score of 3 or 4 was recorded, according to the intensivists' preference.Depending on the sedation regime applied, patients with NIV intolerance are divided into two groups: remifentanil group and dexmedetomidine group.The investigators will compare the two groups with the NIV intolerance score at 15min,1, 3, 6, 12, 24, 48, 60 and 72 hours after the initiation of the sedation regime. The investigators will also compare the two groups with clinical outcomes such as NIV failure, tracheotomy rate, mortality, ICU length of stay etc.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* after cardiac surgery
* receiving noninvasive ventilation
* moderate to severe NIV intolerance (NIV intolerance score of 3 or 4)

Exclusion Criteria:

* difficult expectoration
* pregnancy or breastfeeding
* intensive care delirium screening checklist score more than 4
* drug abuse history
* known allergy to opiods
* cardiogenic shock
* malignant arrhythmias

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult cardiac surgical patients who receive NIV and develop moderate to severe intolerance (NIV intolerance score of 3 or 4) between January 2018 and December 2019 in our CSICU will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guo-wei Tu, PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan hospital, Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Remifentanil Group: Eligible patients will receive a continuous infusion of remifentanil starting with 0.05 μg/kg/min. The doses will be adjusted according to the sedation satisfaction (sedation target is to achieve NIV-intolerance score 1-2), and the maximum dose is 0.12 μg/kg/min.
  Remifentanil: The noninvasive ventilation intolerant patients was sedated by remifentanil.
- Dexmedetomidine Group: Eligible patients will receive a continuous infusion of dexmiditomidine starting with 0.5 μg/kg/h. The doses will be adjusted according to the sedation satisfaction (sedation target is to achieve NIV-intolerance score 1-2), and the maximum dose is 1 μg/kg/h.
  Dexmedetomidine: The noninvasive ventilation intolerant patients was sedated by dexmeditomidine.
Period: Overall Study
Arm/Group | Remifentanil Group | Dexmedetomidine Group
Started | 52 | 38
Completed | 0 | 0
Not Completed | 52 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remifentanil Group | Dexmedetomidine Group | Total
Number analyzed (Participants) | 52 | 38 | 90
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [56 to 73] | 67 [53 to 73] | 65 [54 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 10 | 29
  Male | 33 | 28 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 52 | 38 | 90
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 52 | 38 | 90
baseline NIV intolerance score [Count of Participants; unit: Participants] — In this study, tolerance of NIV is estimated by a four-point NIV intolerance score system: A score of 1 indicates NIV tolerance; a score of 2 indicates mild intolerance with some discomfort and occasional grabbing at the NIV mask; a score of 3 indicates moderate intolerance and discomfort with the NIV mask most of the time with frequent grabbing at the mask (sometimes pulling it off); and a score of 4 indicates severe NIV intolerance with agitation or/and an inability to leave the NIV mask in place. And higher NIV intolerance score is considered worse outcome.
  Participants
    NIV intolerance score of 4 | 21 | 13 | 34
    NIV intolerance score of 3 | 31 | 25 | 56
    NIV intolerance score of 2 | 0 | 0 | 0
    NIV intolerance score of 1 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With NIV Failure
Description: NIV failure was defined by reintubation or death in the course of this study
Time Frame: 72 hours after the initiation of sedation
Population: Summary statistics are expressed as numbers and percentages and compared between groups by Chi-square test.
Measure: Count of Participants; unit: Participants
Arm/Group | Remifentanil Group | Dexmedetomidine Group
Number analyzed (Participants) | 52 | 38
Participants | 10 | 8
Statistical Analysis 1: Comparison: Remifentanil Group vs Dexmedetomidine Group; Summary statistics are expressed as numbers and percentages and compared between groups by Chi-square test; Test type: Other; p = 0.831, Chi-squared

2. Secondary Outcome: Number of Participants With NIV Mitigation
Description: Mitigation was defined by patients who were relieved from the initial intolerant status
Time Frame: 72 hours after the initiation of sedation
Population: The generalized estimating equations approach was employed to analyze changes in the mitigation rate over time between the two groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Remifentanil Group | Dexmedetomidine Group
Number analyzed (Participants) | 52 | 38
Participants | 44 | 31
Statistical Analysis 1: Comparison: Remifentanil Group vs Dexmedetomidine Group; Test type: Other; p = 0.800, Generalized estimating equations

ADVERSE EVENTS:
Time Frame: 72 hours after the initiation of sedation regime
Arm/Group | Remifentanil Group | Dexmedetomidine Group
All-Cause Mortality (participants affected / at risk) | 6/52 | 4/38
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/38
Other Adverse Events (participants affected / at risk) | 0/52 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT03395886/Prot_SAP_000.pdf